CLINICAL TRIAL: NCT05426707
Title: Efficacy and Safety of Remote Ischemic Conditioning for the Treatment of Resistant Hypertension: a Pilot Study
Brief Title: Remote Ischemic Conditioning for the Treatment of Resistant Hypertension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ji Xunming,MD,PhD (Other)
Responsible Party: Sponsor-Investigator, Ji Xunming,MD,PhD, Professor, Capital Medical University
Organization: Capital Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RIC-Resistant HTN
Record Dates: First submitted 2022-06-16; First posted 2022-06-22 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Resistant Hypertension
Keywords: Resistant Hypertension; Remote ischemic conditioning

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RIC group (Experimental): RIC is a non-invasive therapy that is performed by automated pneumatic cuffs placed on bilateral arms. The RIC protocol includes five cycles of 5-min inflation to 200mmHg and 5-min deflation.
  Interventions: Device: RIC
- Sham RIC group (Sham Comparator): The Sham-RIC protocol include five cycles of 5-min inflation to 60 mmHg and 5-min deflation by placing automated pneumatic cuffs on bilateral arms.
  Interventions: Device: Sham-RIC

INTERVENTIONS:
Device: RIC — RIC is a non-invasive therapy that is performed by automated pneumatic cuffs placed on bilateral arms. The RIC protocol includes five cycles of 5-min inflation to 200mmHg and 5-min deflation.
  Arms: RIC group
Device: Sham-RIC — The Sham-RIC protocol include five cycles of 5-min inflation to 60 mmHg and 5-min deflation by placing automated pneumatic cuffs on bilateral arms.
  Arms: Sham RIC group

SUMMARY:
This study aims to explore the efficacy and safety of remote ischemia adaptation for the treatment of resistant hypertension.

DETAILED DESCRIPTION:
Resistant hypertension is defined as a blood pressure of 140/90 mmHg or higher despite adherence to at least three antihypertensive drugs (including one diuretic), accounting for 20% to 30% of patients with hypertension. Compared with patients with well-controlled blood pressure, the cardiovascular risk of resistant hypertension is increased by about 50%. Limb remote ischemic conditioning (LRIC) triggers endogenous protective effects through transient and repeated ischemia in the limb to protect remote tissues and organs. The mechanisms of LRIC involve the regulation of the autonomic nervous system, the release of humoral factors, improvement of vascular endothelial function, and modulation of immune/inflammatory responses, which can antagonize the pathogenesis of hypertension through multiple pathways to lead to a drop in BP theoretically. This theory has been preliminarily confirmed by several small sample-size studies in non-resistant hypertension. This study aims to explore the efficacy and safety of remote ischemia adaptation for the treatment of resistant hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Aged 30~80 years old;

  * Taking ≥ 3 antihypertensive drugs (including one diuretic) for more than 4 weeks regularly;

    * Office blood pressure ≥ 140/90mmhg, and 24 h average blood pressure ≥ 130/80 mmHg;

      * Willing to participate in the study, follow the study protocol, and provide informed consent.

Exclusion Criteria:

* Secondary hypertension;

  * eGFR<45ml/min/1.73m2；

    * Office blood pressure ≥180/110 mmHg, and 24 h average blood pressure ≥ 170/100 mmHg；

      * Hypertensive crisis occurred within 3 months;

        * Type 1 diabetes;

          * Cardiovascular events occurred within 3 months;

            * Atrial fibrillation;

              * Presence of any severe disease that adversely affects the subject or study;

                * Patients with contraindication for remote ischemic conditioning, such as vascular injury, soft tissue injury, orthopedic injury, or arm infection;

                  * Pregnancy, lactation, or planned pregnancy;

                    * Patients not suitable for this trial considered by researchers for other reasons；

                      * Participation in another device or drug trial simultaneously.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
Changes of 24 h average systolic blood pressure | from baseline to 8 weeks
  Changes of 24 h average systolic blood pressure from baseline to 8 weeks

SECONDARY OUTCOMES:
Changes of 24 h average diasolic blood pressure | from baseline to 8 weeks
  Changes of 24 h average diasolic blood pressure from baseline to 8 weeks
Changes of daytime average systolic blood pressure | from baseline to 8 weeks
  Changes of daytime average systolic blood pressure from baseline to 8 weeks
Changes of daytime average diastolic blood pressure | from baseline to 8 weeks
  Changes of daytime average diastolic blood pressure from baseline to 8 weeks
Changes of nighttime average systolic blood pressure | from baseline to 8 weeks
  Changes of nighttime average systolic blood pressure from baseline to 8 weeks
Changes of nighttime average diastolic blood pressure | from baseline to 8 weeks
  Changes of nighttime average diastolic blood pressure from baseline to 8 weeks
Changes of 24 h average heart rate | from baseline to 8 weeks
  Changes of 24 h average heart rate from baseline to 8 weeks
Changes of office systolic blood pressure | from baseline to 8 weeks
  Changes of office systolic blood pressure from baseline to 8 weeks
Changes of office diastolic blood pressure | from baseline to 8 weeks
  Changes of office diastolic blood pressure from baseline to 8 weeks
Changes of home systolic blood pressure | from baseline to 8 weeks
  Changes of home systolic blood pressure from baseline to 8 weeks
Changes of home diastolic blood pressure | from baseline to 8 weeks
  Changes of home diastolic blood pressure from baseline to 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Xunming Ji, MD, PhD, Principal Investigator — Xuanwu Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No